CLINICAL TRIAL: NCT03964727
Title: A Phase 2 Open-Label Study of Sacituzumab Govitecan (IMMU-132) in Subjects With Metastatic Solid Tumors
Brief Title: Study of Sacituzumab Govitecan in Participants With Metastatic Solid Tumors
Acronym: TROPiCS-03
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-11; 2019-000579-18 (EudraCT Number); 2024-513611-28 (Other: European Medicines Agency)
Record Dates: First submitted 2019-04-29; First posted 2019-05-28 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 Group 1: NSCLC [Adenocarcinoma + Squamous Cell Carcinoma (SCC)] (Experimental): Based on protocol amendment 1, participants with non-small cell lung cancer (NSCLC) subtypes such as adenocarcinoma and SCC with high trophoblast cell-surface antigen 2 (Trop-2) expression will receive sacituzumab govitecan-hziy (SG) 10 mg/kg of body weight, administered as a slow intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria will be met.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 1 Group 2: NSCLC (Adenocarcinoma) (Experimental): Based on protocol amendment 2 or 3, participants with NSCLC subtype of adenocarcinoma with or without high Trop-2 expression will receive SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria will be met.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 1 Group 3: NSCLC (SCC) (Experimental): Based on protocol amendment 2 or 3, participants with NSCLC subtype of SCC with or without high Trop-2 expression will receive SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria will be met.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 2: Head And Neck Squamous Cell Carcinoma (HNSCC) (Experimental): Participants with HNSCC will receive SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria will be met.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 3: Endometrial Cancer (EC) (Experimental): Participants with EC will receive SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria will be met.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 4: Extensive-Stage Small Cell Lung Cancer (ES-SCLC) (Experimental): Participants with ES-SCLC will receive SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria will be met.
  Interventions: Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; GS-0132

SUMMARY:
The goal of this clinical study is to learn more about the study drug, sacituzumab govitecan-hziy, in participants with metastatic (cancer that has spread) solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with the following histologically documented metastatic (M1, Stage IV) or locally advanced solid tumors

  * NSCLC [adenocarcinoma or squamous cell carcinoma (SCC)] that has progressed after prior platinum-based chemotherapy and programmed death-(ligand) 1 (PD-(L)1) directed therapy
  * HNSCC that has progressed after prior platinum-based chemotherapy and anti-PD-(L)1 directed therapy No more than 3 prior lines of systemic treatment is allowed
  * Endometrial carcinoma that has progressed after prior platinum-based chemotherapy and anti-PD-(L)1 directed therapy No more than 3 prior lines of systemic treatment is allowed.
  * Extensive stage SCLC that has progressed after prior platinum-based chemotherapy and PD-(L)1 directed therapy. No more than one prior line of systemic treatment is allowed (re-challenge with the same initial regimen is not allowed)
* Eastern Cooperative Oncology Group (ECOG) Performance status score of 0 or 1
* Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation
* Adequate hepatic and renal function [Creatinine Clearance (CrCl) ≥30mL/min]
* Individual must have at least a 3-month life expectancy
* Have measurable disease by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria

Key Exclusion Criteria:

* Have had a prior anti-cancer biologic agent within 4 weeks prior to study Day 1 or have had prior chemotherapy, targeted small molecule therapy, radiation therapy within 2 weeks prior to Study Day 1
* Have not recovered (i.e., ≤ Grade 1) from adverse events due to a previously administered agent
* Have previously received topoisomerase I inhibitors
* Have an active second malignancy
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Individuals with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases and are taking ≤20 mg/day of prednisone or its equivalent. All individuals with carcinomatous meningitis are excluded regardless of clinical stability
* Additional cohort specific exclusion criteria

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (65):
- United States (31):
  - Alaska Oncology & Hematology, LLC, Anchorage, Alaska
  - USOR - Arizona Oncology - Glendale - Saguaro Cancer Center, Glendale, Arizona
  - Arizona Oncology Associates PC-HAL, Goodyear, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - UCLA Hematology/Oncology, Los Angeles, California
  - TRIO-US Central Administration, Whittier, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Smilow Cancer Hospital at Yale, New Haven, Connecticut
  - SIU School of Medicine, Simmons Cancer Institute at SIU, Springfield, Illinois
  - PathGroup Labs, LLC, Fort Wayne, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Christus Highland Cancer Treatment Center, Shreveport, Louisiana
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - North Mississippi Medical Center - Hematology and Oncology - Tupelo, Tupelo, Mississippi
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - David C. Pratt Center, St Louis, Missouri
  - Comprehensive Cancer of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology - Albany Medical Center, Albany, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine - Upper East Side, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Willamette Valley Cancer Institute and Research Center - Eugene, Eugene, Oregon
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Blue Ridge Cancer Care - Wytheville, Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
- Australia (9):
  - Southern Highlands Cancer Center, Bowral, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Blacktown Hospital, Westmead, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Mater Cancer Centre, Mater Misericordiae Limited, South Brisbane, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Monash Medical Centre, Monash Health, Clayton, Victoria
  - The Andrew Love Cancer Centre, Geelong Hospital, Geelong, Victoria
- Belgium (2):
  - Cliniques Universitaires UCL Saint-Luc, Brussels
  - Grand Hopital de Charleroi asbl (GHdC), Charleroi
- Canada (4):
  - Cross Cancer Institute, Edmonton
  - London Health Sciences Centre- Victoria Hospital, London
  - Jewish General Hospital, Montreal
  - The Ottawa Hospital, Ottawa
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre George Francois Leclerc, Dijon
  - Institut Claudius Régaud - IUCT Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Hong Kong (5):
  - Hong Kong Integrated Oncology Centre, Central
  - Hong Kong Sanatorium & Hospital, Happy Valley
  - Queen Mary Hospital, Hong Kong
  - Hong Kong United Oncology Center, Kowloon
  - Department of Clinical Oncology, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Taipei TzuChi Hospital, New Taipei City
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Medical Foundation, Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santin AD, Corr BR, Spira A, Willmott L, Butrynski J, Tse KY, Patel J, Mekan S, Wu T, Lin KW, Kuo P, Dumbrava EE. Efficacy and Safety of Sacituzumab Govitecan in Patients With Advanced Solid Tumors (TROPiCS-03): Analysis in Patients With Advanced Endometrial Cancer. J Clin Oncol. 2024 Oct 10;42(29):3421-3429. doi: 10.1200/JCO.23.02767. Epub 2024 Jul 31. PMID 39083724
- [Background] Michel L, Jimeno A, Sukari A, Beck JT, Chiu J, Ahern E, Hilton J, Even C, Zanetta S, Mekan S, Patel J, Wu T, Dumbrava EE. Sacituzumab Govitecan in Patients with Relapsed/Refractory Advanced Head and Neck Squamous Cell Carcinoma: Results from the Phase II TROPiCS-03 Basket Study. Clin Cancer Res. 2025 Mar 3;31(5):832-838. doi: 10.1158/1078-0432.CCR-24-2523. PMID 39665770
- [Background] Dowlati A, Chiang AC, Cervantes A, Babu S, Hamilton E, Wong SF, Tazbirkova A, Sullivan IG, van Marcke C, Italiano A, Patel J, Mekan S, Wu T, Waqar SN. Phase 2 Open-Label Study of Sacituzumab Govitecan as Second-Line Therapy in Patients With Extensive-Stage SCLC: Results From TROPiCS-03. J Thorac Oncol. 2025 Jun;20(6):799-808. doi: 10.1016/j.jtho.2024.12.028. Epub 2025 Jan 2. PMID 39755168
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=IMMU-132-11

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, France, Australia, Hong Kong, Spain, Taiwan, Canada, and Belgium.
Pre-assignment Details: 396 participants were screened. Data submitted represent primary analysis performed on data collected by the Primary Completion Date. Complete data will be submitted within 1 year of the study completion date.
Groups:
- Cohort 1 Group 1: NSCLC [Adenocarcinoma + Squamous Cell Carcinoma (SCC)]: Based on protocol amendment 1, participants with non-small cell lung cancer (NSCLC) subtypes such as adenocarcinoma and SCC with high trophoblast cell-surface antigen 2 (Trop-2) expression received sacituzumab govitecan-hziy (SG) 10 mg/kg of body weight, administered as a slow intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 22.1 months).
- Cohort 1 Group 2: NSCLC (Adenocarcinoma): Based on protocol amendment 2 or 3, participants with NSCLC subtype of adenocarcinoma with or without high Trop-2 expression received SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 38.7 months).
- Cohort 1 Group 3: NSCLC (SCC): Based on protocol amendment 2 or 3, participants with NSCLC subtype of SCC with or without high Trop-2 expression received SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 20.7 months).
- Cohort 2: Head And Neck Squamous Cell Carcinoma (HNSCC): Participants with HNSCC received SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 12.3 months).
- Cohort 3: Endometrial Cancer (EC): Participants with EC received SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 40.0 months).
- Cohort 4: Extensive-Stage Small Cell Lung Cancer (ES-SCLC): Participants with ES-SCLC received SG 10 mg/kg of body weight, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 29.3 months).
Period: Overall Study
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + Squamous Cell Carcinoma (SCC)] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: Head And Neck Squamous Cell Carcinoma (HNSCC) | Cohort 3: Endometrial Cancer (EC) | Cohort 4: Extensive-Stage Small Cell Lung Cancer (ES-SCLC)
Started | 31 | 34 | 31 | 43 | 41 | 43
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 31 | 34 | 31 | 43 | 41 | 43
Not completed — Death | 14 | 23 | 25 | 31 | 28 | 32
Not completed — Still on study | 0 | 6 | 2 | 4 | 7 | 8
Not completed — Reason not specified | 16 | 3 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 7 | 4 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of SG.
Groups:
- Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC]: Based on protocol amendment 1, participants with NSCLC subtypes such as adenocarcinoma and SCC with high Trop-2 expression received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 22.1 months).
- Cohort 1 Group 2: NSCLC (Adenocarcinoma): Based on protocol amendment 2 or 3, participants with NSCLC subtype of adenocarcinoma with or without high Trop-2 expression received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 38.7 months).
- Cohort 1 Group 3: NSCLC (SCC): Based on protocol amendment 2 or 3, participants with NSCLC subtype of SCC with or without high Trop-2 expression received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 20.7 months).
- Cohort 2: HNSCC: Participants with HNSCC received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 12.3 months).
- Cohort 3: EC: Participants with EC received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 40.0 months).
- Cohort 4: ES-SCLC: Participants with ES-SCLC received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 29.3 months).
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC | Total~(N=223)
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 14 | 32 | 15 | 17 | 110
  >=65 years | 15 | 18 | 17 | 11 | 26 | 26 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8.7) | 64 (10.5) | 65 (8.4) | 61 (6.8) | 66 (9.1) | 66 (8.2) | 64 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 8 | 10 | 41 | 23 | 116
  Male | 16 | 15 | 23 | 33 | 0 | 20 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 2 | 2 | 6
  Not Hispanic or Latino | 30 | 31 | 29 | 40 | 34 | 36 | 200
  Unknown or Not Reported | 1 | 1 | 2 | 3 | 5 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 23 | 26 | 24 | 33 | 21 | 36 | 163
  Race: Black or African American | 6 | 3 | 3 | 1 | 1 | 2 | 16
  Race: Asian | 0 | 5 | 1 | 4 | 8 | 2 | 20
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2 | 0 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Other or More Than One Race | 1 | 0 | 2 | 0 | 3 | 1 | 7
  Race: Unknow or Not Reported | 1 | 0 | 1 | 2 | 6 | 2 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 32 | 26 | 34 | 28 | 22 | 173
  France | 0 | 0 | 3 | 5 | 2 | 2 | 12
  Australia | 0 | 0 | 1 | 1 | 4 | 5 | 11
  Hong Kong | 0 | 2 | 1 | 1 | 5 | 0 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Taiwan | 0 | 0 | 0 | 1 | 1 | 2 | 4
  Canada | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Belgium | 0 | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Investigator's Assessment
Description: ORR was defined as the percentage of participants who had the best overall response of either complete response (CR) or partial response (PR). Responses are based on the investigator-assessed tumor response using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) criteria for each histologic cohort. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; PR: >30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. The ORR rate was calculated with a two-sided exact 95% CI using the Clopper-Pearson method. Percentages are rounded off.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: The Full Analysis Set included all participants who received at least 1 dose of SG.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43
percentage of participants | 12.9 [3.6 to 29.8] | 5.9 [0.7 to 19.7] | 6.5 [0.8 to 21.4] | 16.3 [6.8 to 30.7] | 26.8 [14.2 to 42.9] | 44.2 [29.1 to 60.1]

2. Secondary Outcome: ORR According to RECIST 1.1 by Blinded Independent Central Review (BICR) Assessment
Description: ORR was defined as the percentage of participants who had the best overall response of either CR or PR. Responses are based on BICR assessment using RECIST 1.1 criteria for each histologic cohort. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal; PR: >30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. The ORR rate was calculated with a two-sided exact 95% CI using the Clopper-Pearson method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43
percentage of participants | 3.2 [0.1 to 16.7] | 8.8 [1.9 to 23.7] | 16.1 [5.5 to 33.7] | 18.6 [8.4 to 33.4] | 24.4 [12.4 to 40.3] | 44.2 [29.1 to 60.1]

3. Secondary Outcome: Duration of Response (DOR) According to RECIST 1.1 by BICR Assessment
Description: DOR was the date of the first evaluation showing documented response, either PR or CR, to date of the first progression of disease (PD) or death from any cause,whichever comes first. Response are according to RECIST 1.1 by BICR for each histological cohort. CR: Disappearance of all target and non-target lesions; and normalization of tumor marker levels initially above upper limits of normal;PR: >30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Disease progression was defined as an increase of >20% in the sum of diameters of target lesions, taking as reference the smallest sum on study(this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of more than 5 mm or the appearance of ≥ 1 new non-target lesions and/or unequivocal progression of existing non-target lesions. DOR was estimated using Kaplan-Meier estimate. The 95% CI was computed by Brookmeyer-Crowley method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set who achieved confirmed CR or PR/with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 1 | 3 | 5 | 8 | 10 | 19
months | 2.86 [NA to NA] — Upper and lower limit of confidence interval (CI) were not estimable due to low number of participants with events. | 22.08 [10.55 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 4.70 [2.10 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 8.67 [2.83 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 16.00 [2.76 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 6.01 [2.92 to 10.22]

4. Secondary Outcome: Clinical Benefit Rate (CBR) According to RECIST 1.1 by BICR Assessment
Description: CBR was percentage of participants with best overall response of CR, PR,or durable stable disease (SD) (SD ≥ 6 months after first dose). Responses are according to RECIST 1.1 by BICR.CR: Disappearance of all target and non-target lesions;& normalization of tumor marker levels initially above upper limits of normal;PR:>30% decrease in sum of LD of target lesions, taking as reference the baseline sum LD. SD:Neither sufficient shrinkage for PR nor sufficient increase for PD, taking reference of smallest sum LD since treatment started or ≥ 1 non-target lesions with maintenance of tumor marker level above normal limits.PD: Increase of >20% in sum of diameters of target lesions, taking reference of smallest sum(this includes baseline sum if smallest on study), the sum must also demonstrate an absolute increase of more than 5 mm or of ≥ 1 new non-target lesions and/or unequivocal progression of existing non-target lesions. Two-sided CI was based on Clopper-Pearson method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43
percentage of participants | 29.0 [14.2 to 48.0] | 23.5 [10.7 to 41.2] | 19.4 [7.5 to 37.5] | 27.9 [15.3 to 43.7] | 39.0 [24.2 to 55.5] | 46.5 [31.2 to 62.3]

5. Secondary Outcome: Progression-free Survival (PFS) According to RECIST 1.1 by BICR Assessment
Description: PFS was defined as the time from the first dose until objective tumor progression or death from any cause, whichever comes first. Responses are according to RECIST 1.1 by BICR. Disease progression was defined as an increase of >20% in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of more than 5 mm or the appearance ≥ 1 new non-target lesions and/or unequivocal progression of existing non-target lesions. PFS was estimated using Kaplan-Meier estimate. The 95% CI for median was computed by Brookmeyer-Crowley method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43
months | 4.11 [2.50 to 7.52] | 4.24 [2.27 to 7.59] | 2.73 [1.41 to 5.49] | 3.25 [1.74 to 6.47] | 5.55 [2.79 to 9.59] | 4.40 [3.19 to 6.67]

6. Secondary Outcome: DOR According to RECIST 1.1 by Investigator's Assessment
Description: DOR was the date of the first evaluation showing documented response, either PR or CR, to date of the first PD or death from any cause, whichever comes first. Responses are based on investigator-assessed tumor response by RECIST 1.1 criteria for each histological cohort.CR:Disappearance of all target and non-target lesions;and normalization of tumor marker levels initially above upper limits of normal;PR:>30% decrease in the sum of the LD of target lesions,taking as reference the baseline sum LD. Disease progression was defined as increase of >20% in sum of diameters of target lesions, taking as reference the smallest sum on study(this includes the baseline sum if that is the smallest on study).In addition, the sum must also demonstrate an absolute increase of more than 5 mm or the appearance of ≥ 1 new non-target lesions and/or unequivocal progression of existing non-target lesions. DOR was estimated using Kaplan-Meier estimate. The 95% CI was computed by Brookmeyer-Crowley method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set who achieved confirmed CR or PR/with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 4 | 2 | 2 | 7 | 11 | 19
months | 8.56 [6.41 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 21.09 [11.10 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 7.87 [6.05 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 4.21 [2.60 to 8.67] | 9.92 [2.79 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 6.31 [3.52 to 10.22]

7. Secondary Outcome: CBR According to RECIST 1.1 by Investigator's Assessment
Description: CBR was the percentage of participants with the best overall response of CR, PR,or durable SD (SD ≥ 6 months after first dose) by investigator-assessed tumor response using RECIST 1.1 criteria.CR:Disappearance of all target and non-target lesions;& normalization of tumor marker levels initially above upper limits of normal;PR:>30% decrease in sum of LD of target lesions,taking as reference the baseline sum LD. SD:Neither sufficient shrinkage for PR nor sufficient increase for PD,taking reference of smallest sum LD since treatment started or ≥ 1 non-target lesions with maintenance of tumor marker level above normal limits.PD: Increase of >20% in sum of diameters of target lesions,taking reference of smallest sum(this includes baseline sum if smallest on study),the sum must also demonstrate an absolute increase of more than 5 mm or of ≥ 1 new non-target lesions and/or unequivocal progression of existing non-target lesions.Two-sided CI was based on Clopper-Pearson method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43
percentage of participants | 32.3 [16.7 to 51.4] | 20.6 [8.7 to 37.9] | 16.1 [5.5 to 33.7] | 30.2 [17.2 to 46.1] | 41.5 [26.3 to 57.9] | 48.8 [33.3 to 64.5]

8. Secondary Outcome: PFS According to RECIST 1.1 by Investigator's Assessment
Description: PFS was defined as the time from the first dose until objective tumor progression or death from any cause, whichever comes first. Responses are based on the investigator-assessed tumor response using RECIST 1.1 criteria. Disease progression was defined as an increase of >20% in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of more than 5 mm or the appearance ≥ 1 new non-target lesions and/or unequivocal progression of existing non-target lesions. PFS was estimated using Kaplan-Meier estimate. The 95% CI for median was computed by Brookmeyer-Crowley method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43
months | 2.79 [1.48 to 7.82] | 3.78 [1.41 to 5.65] | 2.56 [1.41 to 5.49] | 4.14 [1.71 to 5.78] | 4.96 [2.76 to 9.82] | 4.40 [3.81 to 6.11]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval from the first dose date of drug to death from any cause. OS was estimated using Kaplan-Meier estimate. The 95% CI for median was computed by Brookmeyer-Crowley method.
Time Frame: Cohort 1: Up to 5.3 years; Cohort 2: Up to 3.4 years; Cohort 3: Up to 3.3 years; Cohort 4: Up to 2.5 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 31 | 34 | 31 | 43 | 41 | 43
months | 14.26 [4.34 to 23.72] | 11.02 [4.24 to 20.47] | 7.29 [5.16 to 10.22] | 8.97 [7.52 to 12.22] | 14.95 [5.88 to 21.42] | 11.73 [6.57 to 14.72]

10. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any AE with an onset date on or after the study drug start date and no later than 30 days after last dose of study drug or the day before initiation of subsequent therapy, whichever comes first.
Time Frame: Up to 7.2 years
Reporting Status: Not Posted, anticipated posting 2027-12

11. Secondary Outcome: Percentage of Participants Experiencing Clinically Significant Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as any value that increased at least 1 toxicity grade from baseline during the treatment-emergent period.
Time Frame: Up to 7.2 years
Reporting Status: Not Posted, anticipated posting 2027-12

12. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Total SN-38
Description: Cmax was defined as the maximum observed concentration of total SN-38 (the active metabolite of sacituzumab Govitecan-hziy). Cycle length=21 days.
Time Frame: Cohort 1: Post dose: Day 1 of Cycles 1,2,3,7,11,17,23,29,35,41,47; Cohort 2: Post dose: Day 1 of Cycles 1,2,3,7,11,17; Cohort 3: Post dose: Day 1 of Cycles 1,2,3,7,11,17,23,29,35,41,47,53; Cohort 4: Post dose: Day 1 of Cycles 1,2,3,7,11,17,23,29
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of SG per protocol & had at least 1 evaluable posttreatment serum concentration of Total SN-38. Participants with available data were analyzed.As all participants were dosed with same dose of SG, the PK analysis for 3 NSCLC cohorts[Cohort 1 Group 1:NSCLC [Adenocarcinoma + SCC],Cohort 1 Group 2:NSCLC(Adenocarcinoma), and Cohort 1 Group 3:NSCLC(SCC)] were combined. The combined PK data was summarized & reported.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Cohort 1: NSCLC: Participants with NSCLC subtypes such as adenocarcinoma and SCC with high Trop-2 expression (based on protocol amendment 1) and with or without high Trop-2 expression (based on protocol amendment 2 or 3) received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 38.7 months).
- Cohort 3: EC: Participants with EC received SG 10 mg/kg, administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 40 months).
Arm/Group | Cohort 1: NSCLC | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 58 | 39 | 39 | 38
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 | 4790 (1170) | 4410 (734) | 4920 (1060) | 4670 (738)
  Cycle 2 Day 1: number analyzed (Participants) | 46 | 36 | 31 | 33
  Cycle 2 Day 1 | 4420 (1010) | 4210 (807) | 4640 (1840) | 4330 (760)
  Cycle 3 Day 1: number analyzed (Participants) | 34 | 25 | 27 | 33
  Cycle 3 Day 1 | 4280 (1420) | 3930 (1080) | 4440 (1130) | 4150 (1040)
  Cycle 7 Day 1: number analyzed (Participants) | 19 | 13 | 20 | 18
  Cycle 7 Day 1 | 4220 (949) | 3750 (1090) | 4430 (915) | 4210 (1160)
  Cycle 11 Day 1: number analyzed (Participants) | 13 | 3 | 15 | 10
  Cycle 11 Day 1 | 4210 (1200) | 4720 (1210) | 4390 (1030) | 4250 (1390)
  Cycle 17 Day 1: number analyzed (Participants) | 7 | 4 | 9 | 4
  Cycle 17 Day 1 | 4620 (849) | 4700 (647) | 4970 (922) | 5510 (783)
  Cycle 23 Day 1: number analyzed (Participants) | 5 | 0 | 5 | 2
  Cycle 23 Day 1 | 5140 (1090) |  | 4880 (1050) | 5420 (912)
  Cycle 29 Day 1: number analyzed (Participants) | 4 | 0 | 4 | 2
  Cycle 29 Day 1 | 4580 (679) |  | 4720 (499) | 5520 (424)
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 0 | 4 | 0
  Cycle 35 Day 1 | 4360 (1100) |  | 4110 (898) |
  Cycle 41 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 41 Day 1 | 5230 (1150) |  | 5450 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 47 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 47 Day 1 | 4260 (1610) |  | 4580 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 53 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 53 Day 1 |  |  | 5210 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |

13. Secondary Outcome: PK Parameter: Cmax of Free SN-38
Description: Cmax was defined as the maximum observed concentration of free SN-38 (the active metabolite of sacituzumab Govitecan-hziy). Cycle length=21 days.
Time Frame: as for outcome 12
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of SG per protocol & had at least 1 evaluable posttreatment serum concentration of Free SN-38. Participants with available data were analyzed. As all participants were dosed with same dose of SG, the PK analysis for the 3 NSCLC cohorts[Cohort 1 Group 1:NSCLC [Adenocarcinoma + SCC],Cohort 1 Group 2:NSCLC(Adenocarcinoma), and Cohort 1 Group 3:NSCLC(SCC)] were combined.The combined PK data was summarized & reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: NSCLC | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 58 | 39 | 39 | 37
ng/mL
  Cycle 1 Day 1 | 65.4 (23.5) | 200 (386) | 94.5 (143) | 78.5 (60.6)
  Cycle 2 Day 1: number analyzed (Participants) | 46 | 35 | 31 | 33
  Cycle 2 Day 1 | 67.0 (40.2) | 94.9 (160) | 70.2 (69.1) | 87.1 (65.8)
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 25 | 27 | 32
  Cycle 3 Day 1 | 107 (277) | 46.8 (17.2) | 62.5 (41.1) | 74.4 (75.9)
  Cycle 7 Day 1: number analyzed (Participants) | 19 | 13 | 20 | 18
  Cycle 7 Day 1 | 64.6 (26.1) | 70.7 (50.1) | 63.8 (57.2) | 78.7 (63.3)
  Cycle 11 Day 1: number analyzed (Participants) | 13 | 3 | 15 | 10
  Cycle 11 Day 1 | 54.6 (11.1) | 57.1 (29.8) | 59.3 (54.0) | 51.6 (25.2)
  Cycle 17 Day 1: number analyzed (Participants) | 7 | 4 | 9 | 4
  Cycle 17 Day 1 | 56.6 (11.0) | 52.1 (18.1) | 73.3 (37.6) | 74.6 (35.2)
  Cycle 23 Day 1: number analyzed (Participants) | 5 | 0 | 5 | 2
  Cycle 23 Day 1 | 72.8 (35.9) |  | 57.3 (21.2) | 53.0 (17.3)
  Cycle 29 Day 1: number analyzed (Participants) | 4 | 0 | 4 | 2
  Cycle 29 Day 1 | 67.0 (23.0) |  | 158 (140) | 170 (138)
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 0 | 4 | 0
  Cycle 35 Day 1 | 69.4 (51.1) |  | 90.4 (81.3) |
  Cycle 41 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 41 Day 1 | 76.1 (32.3) |  | 158 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 47 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 47 Day 1 | 41.9 (8.77) |  | 369 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 53 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 53 Day 1 |  |  | 239 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |

14. Secondary Outcome: PK Parameter: Cmax of Total Antibody
Description: Cmax was defined as the maximum observed concentration of total antibody of SG [hRS7 immunoglobulin (IgG) and hRS7-SN-38]. Cycle length=21 days.
Time Frame: as for outcome 12
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of SG per protocol & had at least 1 evaluable posttreatment serum concentration of Total Antibody. Participants with available data were analyzed. As all participants were dosed with same dose of SG, the PK analysis for 3 NSCLC cohorts[Cohort 1 Group 1:NSCLC [Adenocarcinoma + SCC],Cohort 1 Group 2:NSCLC(Adenocarcinoma), & Cohort 1 Group 3:NSCLC(SCC)] were combined. The combined PK data was summarized & reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: NSCLC | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 57 | 38 | 38 | 38
ng/mL
  Cycle 1 Day 1 | 232000 (79200) | 209000 (54700) | 249000 (77700) | 222000 (49400)
  Cycle 2 Day 1: number analyzed (Participants) | 46 | 35 | 31 | 32
  Cycle 2 Day 1 | 245000 (79700) | 234000 (98700) | 258000 (114000) | 231000 (73000)
  Cycle 3 Day 1: number analyzed (Participants) | 34 | 25 | 28 | 32
  Cycle 3 Day 1 | 260000 (108000) | 234000 (80600) | 294000 (114000) | 240000 (82100)
  Cycle 7 Day 1: number analyzed (Participants) | 19 | 13 | 20 | 18
  Cycle 7 Day 1 | 272000 (139000) | 245000 (108000) | 305000 (116000) | 260000 (107000)
  Cycle 11 Day 1: number analyzed (Participants) | 12 | 3 | 15 | 10
  Cycle 11 Day 1 | 287000 (120000) | 330000 (114000) | 339000 (123000) | 315000 (132000)
  Cycle 17 Day 1: number analyzed (Participants) | 7 | 4 | 9 | 4
  Cycle 17 Day 1 | 313000 (95800) | 369000 (179000) | 338000 (127000) | 380000 (128000)
  Cycle 23 Day 1: number analyzed (Participants) | 5 | 0 | 5 | 2
  Cycle 23 Day 1 | 356000 (145000) |  | 313000 (104000) | 473000 (45300)
  Cycle 29 Day 1: number analyzed (Participants) | 3 | 0 | 3 | 1
  Cycle 29 Day 1 | 227000 (218000) |  | 360000 (108000) | 506000 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated.
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 0 | 4 | 0
  Cycle 35 Day 1 | 304000 (63700) |  | 286000 (137000) |
  Cycle 41 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 41 Day 1 | 282000 (66500) |  | 434000 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 47 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 47 Day 1 | 257000 (47400) |  | 283000 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 53 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 53 Day 1 |  |  | 281000 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |

15. Secondary Outcome: PK Parameter: Ctrough of Total SN-38
Description: Ctrough was defined as concentration at the end of the dosing interval of total SN-38 (the active metabolite of sacituzumab Govitecan-hziy).
  Cycle length=21 days; C=Cohort; D=Day; EOT=End of Treatment; PD=predose; SFU=Safety Follow-up (up to 30 days after EOT date)
Time Frame: C1:PD,D1:Cycles1,2,3,7,11,17,23,29,35,41,47,EOT(Upto 38.7months)&SFU;C2:PD,D1:Cycles1,2,3,7,11,17,EOT(Upto 12.3months)&SFU;C3:PD,D1:Cycles1,2,3,7,11,17,23,29,35,41,47,53,EOT(Upto 40.0months)&SFU;C4:PD,D1:Cycles1,2,3,7,11,17,23,29,EOT(Upto 29.3months)&SFU
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of SG per protocol & had at least 1 evaluable posttreatment serum concentration of Total SN-38. Participants with available data were analyzed. As all participants were dosed with same dose of SG, the PK analysis for 3 NSCLC cohorts [Cohort 1 Group 1:NSCLC [Adenocarcinoma + SCC],Cohort 1 Group 2:NSCLC(Adenocarcinoma), and Cohort 1 Group 3:NSCLC(SCC)] were combined. The combined PK data was summarized & reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: NSCLC | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 85 | 41 | 39 | 37
ng/mL
  Cycle 1 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 2 Day 1: number analyzed (Participants) | 12 | 11 | 14 | 8
  Cycle 2 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 3 Day 1: number analyzed (Participants) | 30 | 17 | 19 | 13
  Cycle 3 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 7 Day 1: number analyzed (Participants) | 16 | 6 | 13 | 9
  Cycle 7 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 11 Day 1: number analyzed (Participants) | 14 | 2 | 11 | 6
  Cycle 11 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 17 Day 1: number analyzed (Participants) | 12 | 3 | 8 | 3
  Cycle 17 Day 1 | 10.1 (4.05) | 9.78 (2.66) | 10.8 (5.27) | 9.69 (3.46)
  Cycle 23 Day 1: number analyzed (Participants) | 6 | 0 | 1 | 2
  Cycle 23 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | 10.1 (2.99)
  Cycle 29 Day 1: number analyzed (Participants) | 4 | 0 | 3 | 1
  Cycle 29 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | 21.0 (24.4) | 6.68 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated.
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 0 | 2 | 0
  Cycle 35 Day 1 | 7.00 (1.78) |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |
  Cycle 41 Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0
  Cycle 41 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | 6.61 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 47 Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0
  Cycle 47 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | 6.12 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 53 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 53 Day 1 |  |  | 7.55 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  EOT: number analyzed (Participants) | 16 | 10 | 12 | 11
  EOT | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  SFU: number analyzed (Participants) | 1 | 9 | 1 | 12
  SFU | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.

16. Secondary Outcome: PK Parameter: Ctrough of Free SN-38
Description: Ctrough was defined as concentration at the end of the dosing interval of free SN-38 (the active metabolite of sacituzumab Govitecan-hziy).
  Cycle length=21 days; C=Cohort; D=Day; EOT=End of Treatment; PD=predose; SFU=Safety Follow-up (up to 30 days after EOT date)
Time Frame: as for outcome 15
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of SG per protocol and had at least 1 evaluable posttreatment serum concentration of Free SN-38. Participants with available data were analyzed. As all participants were dosed with same dose of SG, the PK analysis for 3 NSCLC cohorts [Cohort 1 Group 1:NSCLC [Adenocarcinoma + SCC],Cohort 1 Group 2:NSCLC(Adenocarcinoma), and Cohort 1 Group 3:NSCLC(SCC)] were combined. The combined PK data was summarized & reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: NSCLC | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 85 | 41 | 39 | 37
ng/mL
  Cycle 1 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 6 | 1
  Cycle 2 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 3 Day 1: number analyzed (Participants) | 4 | 1 | 4 | 1
  Cycle 3 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 17
  Cycle 7 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 11 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 10
  Cycle 11 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 17 Day 1: number analyzed (Participants) | 3 | 4 | 1 | 4
  Cycle 17 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 23 Day 1: number analyzed (Participants) | 2 | 0 | 5 | 2
  Cycle 23 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 29 Day 1: number analyzed (Participants) | 6 | 0 | 1 | 1
  Cycle 29 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 0 | 1 | 0
  Cycle 35 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |
  Cycle 41 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 41 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |
  Cycle 47 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 47 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |
  Cycle 53 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 53 Day 1 |  |  | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. |
  EOT: number analyzed (Participants) | 2 | 29 | 1 | 1
  EOT | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  SFU: number analyzed (Participants) | 8 | 9 | 6 | 12
  SFU | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.

17. Secondary Outcome: PK Parameter: Ctrough of Total Antibody
Description: Ctrough was defined as concentration at the end of the dosing interval of total antibody of SG [hRS7 immunoglobulin (IgG) and hRS7-SN-38].
  Cycle length=21 days; C=Cohort; D=Day; EOT=End of Treatment; PD=predose; SFU=Safety Follow-up (up to 30 days after EOT date)
Time Frame: as for outcome 15
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of SG per protocol & had at least 1 evaluable posttreatment serum concentration of Total Antibody. Participants with available data were analyzed. As all participants were dosed with same dose of SG,the PK analysis for 3 NSCLC cohorts[Cohort 1 Group 1:NSCLC [Adenocarcinoma + SCC],Cohort 1 Group 2:NSCLC(Adenocarcinoma), and Cohort 1 Group 3:NSCLC(SCC)] were combined. The combined PK data was summarized & reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1: NSCLC: Participants with NSCLC subtypes such as adenocarcinoma and SCC with high Trop-2 expression (based on protocol amendment 1) and with or without high Trop-2 expression (based on protocol amendment 2 or 3) received SG 10 mg/kg , administered as a slow IV infusion on Days 1 and 8 of a 21-day treatment cycle until progression of disease, unacceptable toxicity, study withdrawal, death, or another treatment discontinuation criteria was met (up to 38.7 months).
Arm/Group | Cohort 1: NSCLC | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 78 | 41 | 35 | 36
ng/mL
  Cycle 1 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation. | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation.
  Cycle 2 Day 1: number analyzed (Participants) | 48 | 35 | 30 | 32
  Cycle 2 Day 1 | 35200 (24900) | 52600 (44300) | 46200 (36100) | 36000 (26500)
  Cycle 3 Day 1: number analyzed (Participants) | 48 | 25 | 31 | 32
  Cycle 3 Day 1 | 79500 (58200) | 69000 (40700) | 73500 (49100) | 59500 (49600)
  Cycle 7 Day 1: number analyzed (Participants) | 28 | 14 | 28 | 17
  Cycle 7 Day 1 | 89600 (80400) | 70200 (51600) | 107000 (60800) | 65200 (44800)
  Cycle 11 Day 1: number analyzed (Participants) | 21 | 3 | 15 | 10
  Cycle 11 Day 1 | 97500 (77400) | 169000 (67700) | 86900 (46800) | 81600 (44300)
  Cycle 17 Day 1: number analyzed (Participants) | 12 | 4 | 9 | 3
  Cycle 17 Day 1 | 126000 (61500) | 124000 (57700) | 104000 (58800) | 107000 (20400)
  Cycle 23 Day 1: number analyzed (Participants) | 10 | 0 | 5 | 2
  Cycle 23 Day 1 | 80700 (56000) |  | 58200 (41700) | 97300 (13800)
  Cycle 29 Day 1: number analyzed (Participants) | 5 | 0 | 4 | 1
  Cycle 29 Day 1 | 83400 (42200) |  | 71100 (4190082800) | 86100 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated.
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 0 | 3 | 0
  Cycle 35 Day 1 | 94800 (17900) |  | 82800 (105000) |
  Cycle 41 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 41 Day 1 | 39200 (51600) |  | 2660 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 47 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 47 Day 1 | 42100 (56200) |  | 2670 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  Cycle 53 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 53 Day 1 |  |  | 77200 (NA) — Since only 1 participant was analyzed, standard deviation cannot be calculated. |
  EOT: number analyzed (Participants) | 44 | 25 | 24 | 20
  EOT | 54800 (43100) | 64600 (51500) | 62100 (43800) | 56300 (36900)
  SFU: number analyzed (Participants) | 7 | 8 | 6 | 10
  SFU | 33000 (33300) | 23800 (23000) | 45800 (28800) | 18900 (20800)

18. Secondary Outcome: Percentage of Participants With Positive Anti-SG Antibodies
Description: Cycle length=21 days; C=Cohort; D=Day; EOT=End of Treatment; PD=predose; SFU=Safety Follow-up (up to 30 days after EOT date)
Time Frame: as for outcome 15
Population: The Immunogenicity Analysis Set included all enrolled participants who received at least 1 dose of SG and had at least 1 evaluable posttreatment anti-SG antibody test result.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
Number analyzed (Participants) | 30 | 33 | 29 | 43 | 41 | 43
percentage of participants | 0 | 3.0 | 3.4 | 4.7 | 2.4 | 4.7

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events: Up to 5.3 years
Description: All-Cause Mortality: The All Enrolled Analysis Set included all participants who were assigned enrollment dates.; Adverse Events: The Safety Analysis Set included all participants who received at least 1 dose of SG.
Arm/Group | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] | Cohort 1 Group 2: NSCLC (Adenocarcinoma) | Cohort 1 Group 3: NSCLC (SCC) | Cohort 2: HNSCC | Cohort 3: EC | Cohort 4: ES-SCLC
All-Cause Mortality (participants affected / at risk) | 26/31 | 27/34 | 28/31 | 35/43 | 30/41 | 32/43
Serious Adverse Events (participants affected / at risk) | 15/31 | 11/34 | 13/31 | 13/43 | 19/41 | 22/43
Other Adverse Events (participants affected / at risk) | 30/31 | 34/34 | 30/31 | 43/43 | 40/41 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] (N=31) | Cohort 1 Group 2: NSCLC (Adenocarcinoma) (N=34) | Cohort 1 Group 3: NSCLC (SCC) (N=31) | Cohort 2: HNSCC (N=43) | Cohort 3: EC (N=41) | Cohort 4: ES-SCLC (N=43)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1 | 7 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myopericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 2 | 0 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 1 | 2 | 2
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2 | 1 | 1 | 2
Septic encephalopathy (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Group 1: NSCLC [Adenocarcinoma + SCC] (N=31) | Cohort 1 Group 2: NSCLC (Adenocarcinoma) (N=34) | Cohort 1 Group 3: NSCLC (SCC) (N=31) | Cohort 2: HNSCC (N=43) | Cohort 3: EC (N=41) | Cohort 4: ES-SCLC (N=43)
Anemia (Blood and lymphatic system disorders) | 9 | 12 | 6 | 13 | 19 | 13
Leukocytosis (Blood and lymphatic system disorders) | 1 | 4 | 1 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 6 | 8 | 5 | 8 | 6 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 4 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 16 | 16 | 15 | 19 | 24 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 2 | 3 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 2 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 4 | 3 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 3 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 2 | 1 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 5 | 3 | 3 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 11 | 13 | 11 | 6 | 15 | 18
Diarrhoea (Gastrointestinal disorders) | 21 | 17 | 15 | 20 | 22 | 33
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 1 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 2 | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 1 | 4 | 2 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 12 | 20 | 12 | 20 | 23 | 17
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 6 | 1 | 3 | 5 | 7
Vomiting (Gastrointestinal disorders) | 7 | 7 | 7 | 15 | 10 | 8
Chest pain (General disorders) | 2 | 1 | 1 | 0 | 1 | 0
Chills (General disorders) | 1 | 3 | 1 | 0 | 1 | 1
Fatigue (General disorders) | 15 | 20 | 18 | 19 | 24 | 27
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 2 | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 4 | 0 | 0 | 1
Oedema (General disorders) | 0 | 2 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 3 | 6 | 4 | 0 | 6 | 5
Peripheral swelling (General disorders) | 0 | 2 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 5 | 3 | 5 | 2
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 1 | 1 | 2
Covid-19 (Infections and infestations) | 0 | 4 | 2 | 5 | 8 | 5
Herpes zoster (Infections and infestations) | 1 | 2 | 1 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 2 | 2 | 7 | 4 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 3 | 0 | 2 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 2 | 4 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 1 | 7 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1 | 5 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 3 | 0 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 2 | 2 | 4 | 2 | 2 | 4
Blood potassium decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 2 | 2 | 5 | 4 | 4
Weight increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 10 | 11 | 11 | 3 | 10
Dehydration (Metabolism and nutrition disorders) | 4 | 7 | 6 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5 | 5 | 6 | 7 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 3 | 5 | 7 | 11 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 3 | 7 | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 5 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 2 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7 | 1 | 7 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 0 | 0 | 4
Dizziness (Nervous system disorders) | 3 | 5 | 5 | 3 | 3 | 6
Dysgeusia (Nervous system disorders) | 1 | 3 | 1 | 1 | 4 | 6
Headache (Nervous system disorders) | 8 | 8 | 5 | 3 | 5 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 5
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 1 | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 1 | 1 | 1 | 2 | 3
Taste disorder (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2 | 1 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 3 | 0 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 2 | 3 | 1 | 2 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 5 | 4 | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 9 | 11 | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2 | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 6 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 22 | 13 | 16 | 17 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 2 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 6 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 3 | 5 | 8 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 2 | 1
Flushing (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 2 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 3 | 1 | 1 | 2
Hypotension (Vascular disorders) | 6 | 4 | 5 | 4 | 1 | 5
Lymphocele (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03964727/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03964727/SAP_001.pdf